CLINICAL TRIAL: NCT06920966
Title: Recovery Optimization Intervention to Reduce the Risk of Injuries in Soccer Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IGOID1
Record Dates: First submitted 2025-03-20; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Muscle Fatigue (C23.888.592.612.612); Athletic Injuries (C26.857.500.124); Recovery of Function (G11.427.698.620); Cryotherapy (E02.095.301.250); Thermotherapy (E02.095.301.750); Soccer (I03.450.642.845.750); Biomarkers (D23.050.301); Thermography (E01.370.350.700.750); Physical Fitness (G11.427.410.698)
Keywords: Muscle Fatigue; Recovery Interventions; Fatigue Reduction; Recovery Optimization; Physical Performance
MeSH Terms: conditions — Athletic Injuries; Hyperthermia

STUDY DESIGN:
Intervention Model Description: This study employs a randomized crossover design to evaluate the effects of different recovery interventions on reducing muscle fatigue and improving performance in football players. The interventions include cold water immersion (CWI), hot water immersion (HWI), no immersion (NI), and thermography-guided immersion (TI).
  Participants are randomly assigned to different intervention sequences, ensuring each participant receives all interventions in a random order. The study is divided into four blocks, each lasting five weeks. During each block, participants undergo one of the recovery interventions.
  Interventions:
  CWI: Five intermittent immersions of 2 minutes each in cold water (11°C). HWI: Continuous immersion of 18 minutes in hot water (38°C). NI: No immersion. TI: Based on thermographic assessments, participants receive either CWI or HWI. Outcome measures include muscle fatigue, performance metrics, biomarker levels, and subjective recovery assessments.
Masking Description: We selected "None (Open Label)" for masking in this study for several reasons:
  Practicality and Feasibility: The interventions (cold and hot water immersions) are easily distinguishable by participants due to their distinct physical sensations, making blinding impractical.
  Transparency and Compliance: An open-label design allows full transparency with participants, enhancing compliance and cooperation as they understand the procedures and potential benefits.
  Ethical Considerations: Providing complete information respects participants' autonomy and their right to make informed decisions about their participation, especially for physical interventions affecting their health.
  Data Collection and Monitoring: The open-label design facilitates easier monitoring and data collection, improving accuracy and reliability without the need for complex blinding procedures.
  Focus on Objective Measures: The study relies on objective measures (thermography, biomarker analysis, performance tests)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cold Water Immersion (CWI) (Experimental): Participants undergo five intermittent immersions of 2 minutes each in cold water (11°C), with 2-minute rest periods in between.
  Interventions: Other: Cold Water Immersion (CWI)
- Hot Water Immersion (HWI) (Experimental): Participants undergo a continuous immersion of 18 minutes in hot water (38°C).
  Interventions: Other: Hot water immersion (HWI)
- No Immersion (NI) (No Intervention): Participants follow the same protocol structure without any immersion.
- Thermography-Guided Immersion (TI) (Experimental): Based on thermographic assessments, participants with a hypothermic profile (decreased temperature) receive hot water immersion, while those with a hyperthermic profile (increased temperature) receive cold water immersion.
  Interventions: Other: Thermography-Guided Immersion (TI)

INTERVENTIONS:
Other: Cold Water Immersion (CWI) — Participants undergo five intermittent immersions of 2 minutes each in cold water (11°C), with 2-minute rest periods in between.
  Other Names: Intermittent Cold Water Immersion (11ºC)
  Arms: Cold Water Immersion (CWI)
Other: Hot water immersion (HWI) — Participants undergo a continuous immersion of 18 minutes in hot water (38°C)
  Other Names: Continuous hot water immersion (38ºC)
  Arms: Hot Water Immersion (HWI)
Other: Thermography-Guided Immersion (TI) — Based on thermographic assessments, participants with a hypothermic profile (decreased temperature) receive hot water immersion, while those with a hyperthermic profile (increased temperature) receive cold water immersion.
  Arms: Thermography-Guided Immersion (TI)

SUMMARY:
The goal of this clinical trial is to evaluate if recovery interventions using cold and hot water immersion can reduce the risk of injuries in amateur soccer players.

The main questions it aims to answer are:

Do cold water immersions reduce muscle fatigue and improve performance more effectively than hot water immersions? What is the optimal timing and duration for these recovery interventions to maximize their effectiveness?

Researchers will compare:

Cold Water Immersion (CWI) Hot Water Immersion (HWI) No Immersion (NI) Thermographic Immersion (TI) based on individual thermal profiles

Participants will:

Undergo thermographic assessments to determine their thermal profiles. Perform physical tests such as isometric strength tests, countermovement jumps (CMJ), and squats with 50% body weight.

Complete wellness questionnaires to assess their subjective recovery and fatigue levels.

Provide blood and urine samples for biomarker analysis. Participate in recovery interventions (CWI, HWI, or TI) based on their assigned group.

ELIGIBILITY:
Inclusion Criteria:

Age: Participants must be adults (18 years or older). Gender: Both male and female participants are eligible. Sport: Participants must be amateur football players. Team Membership: Participants must be members of a football team in the Castilla-La Mancha regional category.

Consent: Participants must provide written informed consent to participate in the study.

Health: Participants must be in good general health, with no chronic illnesses or conditions that would contraindicate participation in physical activity or water immersion.

Exclusion Criteria:

Injury: Participants who have sustained an injury that prevents them from participating in football activities for at least two weeks during any of the study blocks.

Medical Conditions: Participants with medical conditions that contraindicate water immersion (e.g., severe cardiovascular conditions, open wounds, skin infections).

Withdrawal: Participants who choose to withdraw from the study at any point. Non-compliance: Participants who do not comply with the study protocol or fail to attend scheduled sessions.

Pregnancy: Female participants who are pregnant or planning to become pregnant during the study period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Fatigue Reduction: | From pre-intervention to 48 hours post-intervention
  Evaluated through changes in biomarkers such as creatine kinase (CK), lactate dehydrogenase (LDH), and myoglobin levels, measured at multiple time points (pre- and post-intervention).
Countermovement Jump (CMJ) test | From pre-intervention to 48 hours post-intervention.
  Assessed using the countermovement jump (CMJ) test (cm)
Isometric Strenght Test (Hamstrings) | From pre-intervention to 48 hours post-intervention.
  Assessed using isometric strength tests for the hamstrings (N)
Isometric Strenght Test (Adductor) | From pre-intervention to 48 hours post-intervention.
  Assessed using isometric strength tests for the adductors (N)
Squat Performance | From pre-intervention to 48 hours post-intervention.
  Assessed using squat performance with 50% body weight (reps)

SECONDARY OUTCOMES:
Perceived Recovery | At 24 and 48 hours post-intervention.
  Description: Assessed using the Wellness Questionnaire, which includes questions on perceived recovery.
  Unit of Measure: Score on a scale (1-10) Details: Higher scores indicate better perceived recovery.
Stress Levels | At 24 and 48 hours post-intervention.
  Description: Assessed using the Wellness Questionnaire, which includes questions on stress levels.
  Unit of Measure: Score on a scale (1-10) Details: Higher scores indicate higher stress levels.
Fatigue | At 24 and 48 hours post-intervention.
  Description: Assessed using the Wellness Questionnaire, which includes questions on fatigue.
  Unit of Measure: Score on a scale (1-10) Details: Higher scores indicate higher levels of fatigue.
Muscle Soreness | At 24 and 48 hours post-intervention.
  Description: Assessed using the Wellness Questionnaire, which includes questions on muscle soreness.
  Unit of Measure: Score on a scale (1-10) Details: Higher scores indicate higher levels of muscle soreness.
Sleep Quality | At 24 and 48 hours post-intervention.
  Description: Assessed using the Wellness Questionnaire, which includes questions on sleep quality.
  Unit of Measure: Score on a scale (1-10) Details: Higher scores indicate better sleep quality.
Overall Well-Being | At 24 and 48 hours post-intervention.
  Description: Assessed using the Wellness Questionnaire, which includes questions on overall well-being.
  Unit of Measure: Score on a scale (1-10) Details: Higher scores indicate better overall well-being.
Thermographic Assessments | From pre-intervention to 48 hours post-intervention.
  Monitoring skin temperature changes using thermography to evaluate the effectiveness of the recovery interventions.

OTHER OUTCOMES:
Injury Risk Assessment | From baseline (enrollment) to 24 weeks post-intervention.
  Examining the association between recovery interventions and injury risk, based on the incidence of injuries recorded during the study period.
Concentration of 3-Methylhistidine in Urine | From pre-intervention to 48 hours post-intervention.
  Description: Additional analysis of urine samples for markers such as 3-methylhistidine to assess muscle damage and recovery.
  Unit of Measure: Micrograms per liter (µg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Felipe, PhD, Principal Investigator — University of Castilla-La Mancha

IPD SHARING:
Plan to Share IPD: No
We have decided not to share Individual Participant Data (IPD) with other researchers for several reasons:
  Participant Privacy and Confidentiality: Protecting participant privacy is paramount. Sharing IPD, even de-identified, risks re-identification and breaches confidentiality.
  Ethical Considerations: Our study involves sensitive health and performance data. Limiting access ensures responsible and ethical use, preventing misuse or misinterpretation.
  Data Security: Sharing IPD requires robust security measures to prevent unauthorized access and breaches, which are complex and resource-intensive to maintain.
  Informed Consent: Our consent process did not include provisions for sharing IPD with external researchers. Sharing data without explicit consent would violate ethical approval and participant trust.
  Resource Constraints: Managing data sharing requests and providing necessary support to external researchers require significant resources, which we currently lack.

REFERENCES:
- [Background] Lorenzo Calvo J, Alorda-Capo F, Pareja-Galeano H, Jimenez SL. Influence of Nitrate Supplementation on Endurance Cyclic Sports Performance: A Systematic Review. Nutrients. 2020 Jun 17;12(6):1796. doi: 10.3390/nu12061796. PMID 32560317
- [Background] Bestwick-Stevenson T, Toone R, Neupert E, Edwards K, Kluzek S. Assessment of Fatigue and Recovery in Sport: Narrative Review. Int J Sports Med. 2022 Dec;43(14):1151-1162. doi: 10.1055/a-1834-7177. Epub 2022 Apr 25. PMID 35468639